CLINICAL TRIAL: NCT03401606
Title: Dexmedetomidine vs. Remifentanil for Patient and Surgeon Satisfaction in Cataract Surgery Under Controlled Sedation
Brief Title: Controlled Sedation for Cataract Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: a respiratory depression in remifentanyl group
Sponsor: Fundación Universitaria de Ciencias de la Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 516-3847-33
Record Dates: First submitted 2015-12-14; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Failed Conscious Sedation During Procedure
Keywords: sedation; dexmedetomidine; remifentanil; cataract surgery; surgeon satisfaction; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remifentanil (Active Comparator): remifentanil and dexmedetomidine, 0.25 ng/mL, given intravenous, infusion, until surgery finished.
  Interventions: Drug: remifentanil
- Dexmedetomidine (Active Comparator): dexmedetomidine and remifentanil, 0.125 mcg/kg/hour, given intravenous, infusion, until surgery finished
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: remifentanil — remifentanil, 0.25 ng/mL, given intravenous, infusion, until surgery finished
  Arms: Remifentanil
Drug: Dexmedetomidine — dexmedetomidine, 0.125 mcg/kg/hour, given intravenous, infusion, until surgery finished
  Arms: Dexmedetomidine

SUMMARY:
This study evaluates the surgeon and patient´s satisfaction who undergoes cataract surgery using either dexmedetomidine or remifentanil as sedation

DETAILED DESCRIPTION:
This is a double blind, randomized study which evaluates surgeon and patient´s satisfaction whom undergoes cataract surgery. The surgery was done under local anesthesia and sedation.

ELIGIBILITY:
Inclusion Criteria:

* subject has cataract,
* subject older than 18 years,
* local anesthesia and sedation.

Exclusion Criteria:

* general anesthesia,
* history of consumption of sedatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
Surgeon and patient satisfaction | Intraoperative
  It was evaluated with an absolute numerical subjective scale from 1 to 7, where a score of 1 means total dissatisfaction, and 7 complete satisfaction. Scores were evaluated 30 minutes after surgery begun and at the end of the procedure. Results are presented in median and interquartile ranges.

SECONDARY OUTCOMES:
Heart rate | Intraoperative
  Beats per minute (bpm)
Mean arterial pressure | Intraoperative
  Millimeters of mercury (mmHg)
Hemoglobin oxygen saturation | Intraoperative
  Oxygen saturation (%)
Surgery duration | Intraoperative
  Minutes

OTHER OUTCOMES:
Hypotension | Intraoperative
  Systolic blood pressure below 90 mmHg
Respiratory depression | Intraoperative
  Decreased respiratory rate below 10 rpm and desaturation, situation that required intubation
Oxygen desaturation | Intraoperative
  Hemoglobin oxygen saturation below 90%
Internation | Intraoperative
  Inpatient treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luis Muñoz, Md, Study Director — Fundacion universitaria de ciencias de la salud

IPD SHARING:
Plan to Share IPD: No